CLINICAL TRIAL: NCT04736017
Title: Assessing Effects of Auditory Slow Wave Enhancement on Symptoms and Biomarker Levels in Parkinson Disease and Mild Cognitive Impairment: A Randomized, Double-Blind and Placebo- Controlled Crossover Study
Brief Title: Auditory Slow Wave Enhancement in Parkinson Disease and Mild Cognitive Impairment
Acronym: PDMCI-TS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PDMCI-TS
Record Dates: First submitted 2021-01-25; First posted 2021-02-03 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Parkinson Disease; Mild Cognitive Impairment
Keywords: Parkinson Disease; Mild Cognitive Impairment; Excessive Daytime Sleepiness; Sleep; Slow wave sleep; Auditory enhancement; Neurodegeneration; Cognition
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction; Disorders of Excessive Somnolence; Nerve Degeneration

STUDY DESIGN:
Intervention Model Description: The study is a randomized, double-blind, sham-controlled cross-over trial.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum (Experimental): The device records EEG and other biosignals throughout the night and scans these signals for slow waves associated with deep Non-Rapid Eye Movement (NREM) sleep. Upon recognition of such slow waves and fulfilment of other criteria, a tone is played via the headphones to stimulate and enhance slow waves without waking up the patient.
  Interventions: Device: TSB Axo
- Sham (Sham Comparator): Playing no tones during NREM sleep but wearing the device and recording the biosignals over a period of 2 weeks, every night.
  Interventions: Device: TSB Axo

INTERVENTIONS:
Device: TSB Axo — The TSB Axo is a wearable biosignal recording device combined with an auditory stimulation. The device consists of pre-gelled biosignal electrodes, headphones integrated in a headband, and a biosignal processing module.

SUMMARY:
The study aims to assess the efficacy of auditory slow-wave sleep (SWS) enhancement in PD patients and patients with amnestic MCI. Patients will be randomized to two groups: Group 1 will first be treated with auditory stimulation for two weeks and then - after a washout period - switched to two weeks of sham stimulation. Group 2 will first receive sham stimulation for two weeks and then - after a washout period - switch to two weeks of auditory stimulation treatment. The washout period in between will be 2-4 weeks.

DETAILED DESCRIPTION:
The study is a randomized, double-blind, sham-controlled cross-over trial to assess the efficacy of auditory slow-wave sleep (SWS) enhancement in PD patients and patients with amnestic MCI. The screening phase includes entry questionnaires about inclusion/exclusion criteria, sleep quality, chronotype, and handedness, and 1-4 screening nights at home with the TSB Axo, to allow for stimulation optimization. One of the screening nights will be extended to screen for sleep apnea and periodic limb movements during sleep using an ambulatory screening device. Upon final inclusion, 24 PD and 24 MCI patients will be enrolled in the study for an overall period of 6-8 weeks (not including screening phase). Patients will receive 2 weeks of auditory SWS enhancement and 2 weeks of sham stimulation (only device application, no tones played) in a counter-balanced cross-over design, with a 2-4 week washout period during cross-over. Study visits will be performed immediately before and after each intervention period, i.e. after 2 weeks of auditory stimulation or sham stimulation, respectively. Study visits will include standardized clinical examinations, symptom questionnaires, blood sampling after intervention and screening for adverse events by a study physician. Study visits will take place at the Department of Neurology, University Hospital Zurich.

ELIGIBILITY:
Inclusion Criteria:

* PD: Diagnosis of PD along international criteria, with mild to moderate disease severity (Hoehn and Yahr scale, stages ll-lll)
* PD: Ability to apply the intervention for the duration of study
* MCI: Diagnosis of MCI along international criteria, with a predominant amnestic presentation (single- or multi-domain amnestic MCI)
* MCI: Presence of a cohabitant person who could assist with the application
* MCI: Ability to apply the intervention for the duration of study, with assistance of co-habitant if needed

PD and MCI:

* Age above 18 years
* Informed consent as documented by signature
* Stable home situation (e.g. long-term place to live) that allows for reliable application of intervention for the duration of the study
* Sufficient German language comprehension to follow the study procedures and answer all questions related to the study outcomes
* Dosing of dopaminergic, cholinergic, and other PD or MCI medication must have been stable for at least 14 days prior to start of the first intervention
* Negative pregnancy test during screening (except in women who are surgically sterilized/hysterectomized or postmenopausal for longer than 1 year)

Exclusion Criteria:

* PD: Presence of neurologic, psychiatric, or sleep disorders (others than associated with PD)
* PD: Parkinsonism without response to levodopa; Atypical Parkinsonian syndromes
* PD: Cognitive impairment (Montréal Cognitive Assessment [MoCA] <24)
* MCI: Present diagnosis of a neurological (other than MCI) or interfering psychiatric disease or sleep disorder (e.g. sleep apnoea syndrome, restless legs syndrome)

PD and MCI:

* Severe medical conditions as renal insufficiency, liver failure or congestive heart failure
* Regular use of the following drugs: Benzodiazepines and other central nervous system (CNS)-depressant substances, melatonin and other sleep inducing substances, approved drugs for Alzheimer-type dementia (acetylcholine-esterase inhibitor, memantine)
* Inability to hear the tones produced by the TSB Axo
* Skin disorders/problems/allergies in face/ear area that could worsen with electrode application
* Known or suspected drug- or medication abuse
* Known or suspected non-compliance
* Participation in another study with investigational drug or investigational medical devices within the 30 days preceding and during the present study
* Previous enrolment in the current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Shift work (work during the night)
* Travelling more than 2 time zones in the last month before intervention starts or during intervention (start of intervention will be adapted to fit with this criteria)
* Substance or alcohol abuse (i.e. > 0.5 l wine or 1 l beer per day)
* High caffeine consumption (> 5 servings/day; including coffee, energy drink)
* Implanted deep brain stimulation electrodes
* Women who are pregnant or breast feeding
* Intention to become pregnant during the course of the study
* Lack of safe contraception, defined as: Female patients of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Difference in objective EDS | assessed after each intervention (day 15 of each intervention)
  Difference in objective excessive daytime sleepiness (EDS), measured with Multiple Sleep Latency Test (MSLT; minutes), in Parkinson patients
Difference in verbal episodic memory performance | assessed after each intervention (day 15 of each intervention)
  Difference in verbal episodic memory performance, measured with the Hopkins Verbal Learning Test (HVLT; score ranges from 0 to 12, higher scores indicate better performance) delayed recall, in Mild Cognitive Impairment patients

SECONDARY OUTCOMES:
Subjective EDS | assessed before and after each intervention (day 1 and 15 of each intervention)
  Change in subjective excessive daytime sleepiness (EDS), measured with the Epworth Sleepiness Scale (ESS; score ranges from 0 to 24, higher scores indicate greater EDS)
Sustained attention | assessed after each intervention (day 15 of each intervention)
  Sustained attention, measured with the Sustained Attention to Response Task (SART)
Vigilance | assessed after each intervention (day 15 of each intervention)
  Vigilance, measured with the Psychomotor Vigilance Task (PVT)
Subjective nocturnal sleep quality | assessed before and after each intervention (day 1 and 15 of each intervention)
  Subjective nocturnal sleep quality, measured with the Parkinson's Disease Sleep Scale -2 (PDSS-2; score ranges from 0 to 60, higher scores indicate worse sleep quality) in PD patients and Pittsburgh Sleep Quality Index (PSQI; score ranges from 0 to 21, higher scores indicate worse sleep quality) in MCI patients
Executive Function and attention | assessed after each intervention (day 15 of each intervention)
  Executive function (mental flexibility, verbal fluency, motor programming, sensitivity to interference, working memory, psychomotor processing speed), measured with the Trail Making Test (TMT; in seconds) B/A, the Regensburger Wortflüssigkeitstest (RWT; phonematic and semantic verbal fluency; in word count), the Luria's motor sequence test, the Victoria Stroop Task, the 2-back task, and the TMT A
Plasma biomarkers | assessed after each intervention (day 15 of each intervention)
  Plasma levels of protein accumulation (aSyn, beta-amyloid 40 and 42 [Aß40, Aß40], tau, phosphorylated tau [p-tau]), neurodegeneration (neurofilament light chain; NFL), and synaptic and inflammatory markers
Subjective sleep quality | assessed every morning during the intervention period (days 1-15 of each intervention)
  Subjective sleep quality measured with a Visual Analog Scale (VAS) on a scale from very poor to very good
Subjective mood | assessed every evening during the intervention period (days 1-14 of each intervention)
  Subjective mood during daytime measured with a Visual Analog Scale (VAS) on a scale from very poor to very good
Subjective momentary sleepiness | assessed every evening during the intervention period (days 1-14 of each intervention)
  Subjective momentary sleepiness measured with Karolinska Sleepiness Scale (KSS; score ranges from 1 to 9, higher scores indicate greater momentary sleepiness)
Digital biomarkers | assessed every day during the intervention (days 1-15 of each intervention)
  tapping behavior on tablet
Sleep intensity | assessed continuously during the intervention period (days 1-15 of each intervention)
  Sleep intensity, represented by Slow Wave Activity/ Slow Wave Energy (SWA/SWE), calculated from EEG recordings obtained every night at home with a frontal EEG electrode of the TSB Axo
Depressive symptoms | assessed before and after each intervention (day 1 and 15 of each intervention)
  Depressive symptoms, indicated by the Hospital Anxiety and Depression Scale (HADS; score ranges from 0 to 21, higher scores indicate more depressive symptoms), in MCI patients
Verbal episodic and visuospatial memory function | assessed after each intervention (day 15 of each intervention)
  Verbal episodic and visuospatial memory function, measured with the Hopkins Verbal Learning Test (HVLT; score ranges from 0 to 12, higher scores indicate better performance), and Brief Visuospatial Memory Test (BVMT; score ranges from 0 to 12, higher scores indicate better performance), in MCI patients
Quality of life (VAS) | assessed before and after each intervention (day 1 and 14, day 29 and 42)
  Quality of life, measured with a Visual Analog Scale (VAS) on a scale from very poor to very good, in Parkinson patients
Motor symptoms | assessed before and after each intervention, in the morning prior to dopaminergic medication intake (day 1 and 14 of each intervention)
  Motor symptoms, assessed with the Unified Parkinson's Disease Rating Scale (UPDRS) lll remote version (on tablet; score ranges from 0 to 104, higher scores indicate worse motor symptoms), in Parkinson patients
Focused motor assessment | assessed on day 4 of each intervention
  Assessment of hand/finger movements, in Parkinson patients
Overnight memory consolidation | assessed in the evening of day 13 and in the morning of day 14
  Overnight memory consolidation, assessed with a word-pair task and finger tapping sequence test in PD and MCI patients
Overnight restoration inhibitory control | assessed in the evening of day 13 and in the morning of day 14
  Overnight restoration of inhibitory control, assessed with the Go/NoGo Task (GNG) in PD and MCI patients
Overnight restoration working memory | assessed in the evening of day 13 and in the morning of day 14
  Overnight restoration of the working memory, assessed by the 2-back task in PD and MCI patients
Overnight restoration vigilance | assessed in the evening of day 13 and in the morning of day 14
  Overnight restoration of vigilance, assessed by the Psychomotor Vigilance Test (PVT) in PD and MCI patients

CONTACTS AND LOCATIONS:
Overall Officials: Angelina Maric, PhD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Neurology department, Zurich, Switzerland